CLINICAL TRIAL: NCT06694155
Title: Whey Protein Ingestion and Glucose Control in Pre- and Post Diabetic Individuals
Acronym: DAIRY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Dairy Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 297495
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Prediabetes / Type 2 Diabetes
Keywords: Whey Protein; type II diabetes; Protein turnover; Dietary intake
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The study will enroll 20 prediabetic (A1C 5.7%-6.4%) and 20 diabetic (A1C 6.5%-7.5%) subjects, 50-70 yrs of age, in randomized, crossover fashion. Each subject will participate in two 7d studies, with and without Whey Protein ingestion. Study order will be randomized. Subjects will consume their habitual diets (recorded by dietary log), with the dietary intervention being the additional consumption of two 30g doses of whey on the treatment assignment. Thirty grams of whey or placebo will be ingested within 1hr of waking and prior to breakfast, and a second 30g dose of WPI will be consumed 30min prior to the dinner meal. Main outcomes will be Matsuda index, 24hr glucose AUC, dietary intake (total kcal and macronutrients), and whole-body protein balance. The Matsuda index utilizes an oral glucose tolerance test to derive insulin sensitivity as assessed by euglycemic insulin clamp. Secondary outcomes will be satiety, satiation, and appetite score.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whey Protein Supplementation (Experimental): Crossover study
  Interventions: Dietary Supplement: Whey Protein Isolate Crossover
- Placebo Supplementation (Placebo Comparator): Crossover study
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Whey Protein Isolate Crossover — This crossover intervention includes 1 week of whey protein isolate supplementation and 1 week of placebo supplementation.
  Arms: Whey Protein Supplementation
Dietary Supplement: Placebo — 1 week of Non-whey protein Placebo supplement
  Arms: Placebo Supplementation

SUMMARY:
To examine the effects of twice daily whey protein consumption on blood glucose and insulin in pre-diabetic and diabetic individuals

DETAILED DESCRIPTION:
Protein consumption in the morning has been shown to reduce appetite and caloric intake (19). In addition, premeal whey consumption reduces post prandial blood glucose, reduces gastric emptying rate, and increases peak blood insulin (10). Thus, it is proposed that ingestion of whey protein within 1hr of waking (and prior to breakfast) and 30 minutes prior to dinner will be more effective in suppressing appetite, carbohydrate intake, and glucose AUC. Ingestion upon waking will mitigate the cortisol-induced drive for carbohydrate intake. Ingestion prior to dinner, the most frequently consumed and largest meal in America (20), will reduce food intake, post meal blood glucose, and insulin area under the curve (21).

Specific Aims

1. Determine the effect of WP ingestion within 1hr of waking and prior to breakfast, and 30min prior to dinner, on appetite suppression, carbohydrate and caloric intake, and 24hr glucose AUC over 7d in pre-diabetic (A1C 5.7%-6.4%) and diabetic (A1C 6.5%-7.5%) individuals.
2. Determine the effect of WP ingestion within 1hr of waking and 30min prior to dinner on changes in OGTT, Matsuda index, and whole-body protein balance (compared to control) before and after 7d of WP consumption in pre-diabetic and diabetic individuals.
3. Determine outcome differences between pre-diabetic and diabetic individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ages 50-70 years.
2. Capable of providing informed consent.
3. COVID-19 negative and/or asymptomatic.
4. Willing to abstain from drinking alcohol or consuming marijuana and CBD products during the 7-day study meal period on two occasions.
5. HbA1c: 5.7-6.4% or 6.5% to 7.5%

Exclusion Criteria:

1. Subject who does not/will not eat dairy protein sources.
2. Subjects taking exogenous insulin injections or GLP /GIP injections or other appetite suppressants.
3. Unwilling to keep a detailed 7 day food journal on two occasions
4. Unwilling to wear a CGM for 7 days on two occasions and share the data with the research team.
5. Lactose intolerance.
6. Hemoglobin <10g/dL at screening.
7. History of chemotherapy or radiation therapy for cancer in the 6 months prior to enrollment.
8. History of gastrointestinal bypass/reduction surgery.
9. Pregnant or lactating individuals.
10. History of a chronic inflammatory disease (e.g. Lupus, Crohn's disease)
11. Currently receiving androgen (e.g., testosterone) or anabolic (e.g., GH, IGF-I) therapy.
12. Currently using corticosteroid medications (cortisone, hydrocortisone, prednisone, etc.).
13. Unwilling to avoid using protein or amino-acid supplements during participation.
14. Unwilling to fast overnight.
15. Any medical condition or medication that the PI or clinical study staff finds contradictory to this study.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Whole body protein turnover | 7 days
  Whole body protein turnover reflects the continual synthesis and breakdown of body proteins. It can be measured at a whole-body or tissue level using stable isotope methods.
Oral Glucose Tolerance Test | 7 days
  Oral Glucose Tolerance Test (OGTT) is used to screen for or diagnose diabetes. Normal blood values for a 75 gram OGTT are: Fasting -- 60 to 99 mg/dL (3.3 to 5.5 mmol/L), 1 hour -- Less than 200 mg/dL (11.1 mmol/L), 2 hours -- Less than 140 mg/dL (7.8 mmol/L) is normal.
Blood glucose | 7 days
  Continuous glucose monitoring means using a device to automatically estimate your blood glucose level, also called blood sugar, throughout the day and night for 7 days.

SECONDARY OUTCOMES:
Composite Appetite Scale | 7 days
  A composite appetite scale is a measure used to assess appetite control and influence energy intake. It can be calculated based on factors such as hunger, desire to eat, and fullness rating.
  Appetite Scale:
  How Hungry do you feel? Not Hungry at all <---> Have never been more Hungry How Satisfied do you feel? Completely empty <----> Can't eat another bite How Full do you feel? Not full at all <----> Totally full The more a person is satisfied and feels full and less hungry, the better the outcome is for whey vs placebo supplementation.
Dietary Intake Log | 7 days
  A dietary intake log, also known as a food diary, is a self-reported account of all foods and beverages consumed within a specific timeframe.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Undecided